CLINICAL TRIAL: NCT01137032
Title: An Open -Label Study to Evaluate the Effect of Pandel Cream 0.1% on the Hypothalamic Pituitary Adrenal Axis in the Pediatric and Adult Population
Brief Title: Study to Evaluate Effect of Pandel Cream 0.1% on HPA Axis in Pediatric and Adult Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fougera Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT 0153-01-1
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2016-03-29 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Psoriasis; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pandel Cream 0.1% (Experimental): Pandel Cream 0.1%
  Interventions: Drug: Pandel Cream 0.1%

INTERVENTIONS:
Drug: Pandel Cream 0.1% — A thin coat of cream will be applied and rubbed into the affected areas, as well as normal skin, twice daily for 21 days

SUMMARY:
The purpose of this study is to determine the effect of Pandel® (hydrocortisone probutate cream) Cream 0.1% on the Hypothalamic Pituitary Adrenal (HPA) axis in pediatric and adult subjects with either psoriasis or atopic dermatitis involving greater than 20% body surface area.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis or atopic dermatitis involving more than 20% of body surface area
* Good health with the exception of psoriasis or atopic dermatitis

Exclusion Criteria:

* Any disease affecting the HPA-axis
* Subjects who are pregnant, nursing, or planning a pregnancy within the study participation period

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela C Kaplan, Study Director — Fougera Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Christopher Huerter, MD, Omaha, Nebraska
  - Oswald Mikell, MD, Hilton Head Island, South Carolina
  - Michael Gold, MD, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pandel Cream 0.1%
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pandel Cream 0.1%
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 48.3 [23 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Post-injection Serum Cortisol Level
Description: The number of subjects with a post-injection serum cortisol level less than or equal to 18 ug/dL on Day 22.
Time Frame: 22 Days
Population: 15 subjects represents the subgroup utilized for the analysis of this endpoint.
Measure: Number; unit: participants
Arm/Group | Pandel Cream 0.1%
Number analyzed (Participants) | 15
participants | 1

2. Secondary Outcome: Pre-injection Serum Cortisol Levels
Description: The number of subjects with pre-injection serum cortisol levels less than or equal to 5 ug/dL Day 22.
Time Frame: 22 Days
Population: 15 subjects represents the subgroup utilized for the analysis of this endpoint.
Measure: Number; unit: participants
Arm/Group | Pandel Cream 0.1%
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: and the Number of Subjects With an Increment Between Basal and 30 Minutes Day 22 of at Least 7 ug/dL.
Time Frame: 22 days
Population: 15 subjects represents the subgroup utilized for the analysis of this endpoint.
Measure: Number; unit: participants
Arm/Group | Pandel Cream 0.1%
Number analyzed (Participants) | 15
participants | 1

ADVERSE EVENTS:
Arm/Group | Pandel Cream 0.1%
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 7/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pandel Cream 0.1% (N=19)
PYREXIA (General disorders) | 1
NASOPHARYNGITIS (Infections and infestations) | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
HEADACHE (Nervous system disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
APPLICATION SITE IRRITATION (Skin and subcutaneous tissue disorders) | 1
EAR INFECTION (Infections and infestations) | 1
ANXIETY (Psychiatric disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
DIZZINESS (Nervous system disorders) | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1
OCCULT BLOOD (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other